CLINICAL TRIAL: NCT02803801
Title: Build Your Parenting Toolkit: Guiding Children to Become Flexible Thinkers. SCRC/LIFE Program Pilot Project
Brief Title: Build Your Parenting Toolkit: Guiding Children to Become Flexible Thinkers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehabilitation Centre for Children, Canada (Other)
Responsible Party: Principal Investigator, Lianne Belton, Occupational Therapist, Specialized Communication Resources for Children, Rehabilitation Centre for Children, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BYPT2016
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2017-04-12 (Actual); Status verified 2017-04

CONDITIONS: Autism Spectrum Disorder (ASD); Developmental Disorder
Keywords: Parents' ability to guide their child; Parent perception of competence; Parent understanding of their child's unique learning style
MeSH Terms: conditions — Autism Spectrum Disorder; Developmental Disabilities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Build Your Parenting Toolkit Program (Experimental): Ten session program, with a mix of parents-only lectures and parent and child Cooking Clubs.
  Interventions: Behavioral: Build Your Parenting Toolkit Program

INTERVENTIONS:
Behavioral: Build Your Parenting Toolkit Program — Ten session program, with a mix of parents-only lectures and parent and child Cooking Clubs.

SUMMARY:
This pilot project is a cooperative effort between the Leisure in Fun Environments (LIFE) Program and the Specialized Communication Resources for Children (SCRC) Program at the Rehabilitation Centre for Children (RCC). The investigators will blend and enhance two pre-existing programs in order to provide a new, specialized program for parents of children with ASD or developmental delay. The two programs that will be blended together are "Promoting Flexible Thinking and Interaction with Your Child at Home" and "Saturday Cooking Club." This new program will be a series of ten workshops that alternates between "parents only" learning sessions and practical "cooking club" sessions that allow parents to focus on practicing what they are learning with their child. These programs are based on the principles of Relationship Development Intervention (RDI®), which focuses on providing opportunities to establish a guided participation relationship, which will lead to development of dynamic intelligence and important social thinking abilities. The program is individualized to each child and builds on the principles of typical development to assist the child in achieving social competence. Using this program, children are expected to develop sociability in a naturally progressing order of complexity.

DETAILED DESCRIPTION:
Parenting children with developmental disabilities or Autism Spectrum Disorder (ASD) can be challenging. Often, these children process information in an atypical manner and they may struggle to learn through social engagement. At times, regular parenting techniques do not work with these children, which may leave parents feeling distressed and confused. In their ground breaking interpretation of the International Classification of Functioning, Health and Disability (ICF), The 'F-words' in childhood disability, (2011) Dr. P. Rosenbaum and Dr. J. Gorter state that, "Family represents the essential environment of all children." They point to research that confirms that parental physical and mental health is challenged in families who have a child with a disability. Specifically, behavioural issues of these children significantly contribute to parental stress scores, impact attachment, the relationship with a spouse, parental depression and in particular, a sense of competence. By providing parents the opportunity to understand their child's unique learning style, and the opportunity to learn how to mindfully engage their child, it is the investigators' goal to restore parental competence and the natural parent/child relationship.

The objectives of this new learning series program are to help parents understand their child's unique learning style and to give parents the practical tools to become their child's best teacher and guide. Becoming a mindful parent requires a solid understanding of the child's underlying social learning challenges, and it requires parents to be both self-reflective and analytical. Behaviour change takes time and repeated experience. Parents also need the opportunity to practice in a safe and supportive environment. This learning series will consist of ten in-person sessions, over a period of 12-14 weeks.

ELIGIBILITY:
Inclusion criteria:

- parents of children who have high functioning Autism Spectrum Disorder or high functioning developmental delay, and are aged 7-12

Exclusion criteria:

- unable to complete the study sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-09; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Relationship Development Assessment | 14 weeks
  Video recordings of the parent and child cooking, used to evaluate the parents' responsiveness, communication and ability to stage engagements with their own child
Being a Parent Scale | 14 weeks
  This short questionnaire evaluates parent's current perceptions of a variety of common parenting situations and their emotional reactions

SECONDARY OUTCOMES:
Cooking Club Feedback Questionnaires | 14 weeks
  These questionnaires will be used to evaluate whether the lecture sessions adequately prepared them for the related Cooking Club. These questionnaires will also help parents develop goals to work on at home.
Exit Questionnaire | 14 weeks
  Satisfaction questionnaire, to help improve the program in the future.

CONTACTS AND LOCATIONS:
Overall Officials: Lianne Belton, OT, Principal Investigator — Rehabilitation Centre for Children; Carol Kehler, PT, Principal Investigator — Rehabilitation Centre for Children
Locations (1):
- Rehabilitation Centre for Children, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No